CLINICAL TRIAL: NCT04387201
Title: GLP-1 Therapy: The Role of IL-6 Signaling and Adipose Tissue Remodeling in Metabolic Response
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Absalon D Gutierrez, Associate Professor of Medicine, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-MS-19-0787; R21DK122234 (NIH)
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Glucose Intolerance; Overweight and Obesity; Drug Effect; Adiposity
Keywords: GLP-1; prediabetes; brown fat; adipose tissue; IL-6
MeSH Terms: conditions — Glucose Intolerance; Overweight; Obesity; Prediabetic State | interventions — Vitamin B 12; dulaglutide

STUDY DESIGN:
Intervention Model Description: Crossover clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyanocobalamin, then Dulaglutide (Experimental): Participants first received Cyanocobalamin (vitamin B12) 1000 mcg subcutaneous weekly for 6 weeks. After a washout period of 3 weeks, they then received Dulaglutide 0.75 mg subcutaneous weekly for 2 weeks, followed by 1.5 mg subcutaneous weekly for 4 weeks
  Interventions: Drug: Cyanocobalamin; Drug: Dulaglutide
- Dulaglutide, then Cyanocobalamin (Experimental): Participants first received Dulaglutide 0.75 mg subcutaneous weekly for 2 weeks, followed by 1.5 mg subcutaneous weekly for 4 weeks. After a washout period of of 3 weeks, they then Cyanocobalamin (vitamin B12) 1000 mcg subcutaneous weekly for 6 weeks.
  Interventions: Drug: Cyanocobalamin; Drug: Dulaglutide

INTERVENTIONS:
Drug: Cyanocobalamin — Cyanocobalamin (vitamin B12) 1000 mcg subcutaneous weekly for 6 weeks.
  Other Names: Vitamin B12
Drug: Dulaglutide — Dulaglutide 0.75 mg subcutaneous weekly for 2 weeks, followed by 1.5 mg subcutaneous weekly for 4 weeks
  Other Names: Trulicity

SUMMARY:
This project investigates the anti-obesity mechanisms of glucagon-like peptide-1 (GLP-1) analogs, which are used in the treatment of human obesity and diabetes mellitus. The investigators will test if GLP-1 induces secretion of interleukin-6 (IL-6), a cytokine that may collaborate with GLP-1 analogs to induce the formation of brown fat, which has anti-diabetic properties. The results will guide future obesity and diabetes mellitus therapies.

DETAILED DESCRIPTION:
Incretins, the analogs of glucagon-like peptide-1 (GLP-1), improve glucose control in type 2 diabetes mellitus and counteract obesity through mechanisms that are not completely understood. The investigators' preliminary data show that, in prediabetic human subjects and mice, GLP-1 analog therapy induces an increase in plasma interleukin-6 (IL-6), a cytokine activating signal transducer and activator of transcription 3 (STAT3) signaling, which induces brown (beige) adipocyte differentiation in adipose tissue (AT). The investigators discovered that plasma IL-6 induction occurs through GLP-1 receptor (GLP-1R) stimulation in leukocytes. Interestingly, studies in rodents indicate that GLP-1 / GLP-1R signaling also induces AT beiging. Based on these observations, the investigators hypothesize that incretins induce AT browning in part via transient IL-6 / IL-6 receptor (IL-6R) / STAT3 signaling. The primary objective is to further elucidate the role of IL-6 and GLP-1 signaling in mediating beneficial metabolic effects of incretin therapy. Studies will be paralleled in a human clinical trial, a human cell culture model, and a mouse diet-induced obesity model. GLP-1 analog therapy combined with an IL-6 blocking antibody will be used. Specific Aim 1 is to (A) investigate IL-6 induction / downstream STAT3 signaling and AT browning upon incretin therapy in prediabetic human subjects; and (B) validate mice as a model to study incretin-induced IL-6 signaling as a mediator of AT browning. Specific Aim 2 is to (A) investigate if GLP-1 analog effects on beige adipogenesis depend on IL-6 signaling in human adipocyte progenitors; and (B) investigate if GLP-1 analog effects on beige adipogenesis depend on IL-6 signaling in mice. It is expected that 1) GLP-1 analog signaling via GLP-1R induces IL-6 secretion by leukocytes, and 2) GLP-1 analog therapy induces adipose tissue browning via both direct GLP-1 / GLP-1R signaling and indirect incretin-induced IL-6 / IL-6R / STAT3 signaling. The results of this novel study will give critical insights on the anti-obesity mechanisms of GLP-1 analogs and serve as the basis for developing more targeted therapies for diabetes and obesity. Understanding the anti-diabetic IL-6 effects will also be important for interpreting the results of IL-6 blockade, a therapeutic approach for patients with diabetes and other inflammatory conditions, which may need to be re-considered.

ELIGIBILITY:
Inclusion criteria:

1. Men and women, ages 18-50 years
2. Diagnosis of Prediabetes - defined as either impaired fasting glucose (fasting glucose of 100-125 mg/dL), impaired glucose tolerance (2-hour postprandial blood glucose of 140-199 mg/dL after 75-gram oral glucose challenge), and/or a hemoglobin A1C ranging from 5.5% to 6.4%.
3. BMI ≤ 35 kg/m2
4. Women of childbearing age must agree to use an acceptable method of pregnancy prevention (barrier methods, abstinence, oral contraception, vaginal rings, long-acting reversible contraceptives, or surgical sterilization) for the duration of the study
5. Patients must have the following laboratory values: Hematocrit ≥ 33 vol%, estimated glomerular filtration rate ≥ 60 mL/min per 1.73 m2, AST (SGOT) < 2.5 times ULN, ALT (SGPT) < 2.5 times ULN, alkaline phosphatase < 2.5 times ULN
6. If patients are receiving antihypertensive medications (other than beta blockers) and/or lipid-lowering medications, they must remain on stable doses for the duration of the study.
7. If patients are receiving NSAIDs or antioxidant vitamins, these must be discontinued one week prior to study initiation and cannot be restarted during the study.
8. If patient takes thyroid medications, these must be dosed to control hypo- or hyperthyroidism.

Exclusion Criteria:

1. History of Type 1 or Type 2 diabetes mellitus
2. Pregnant or breastfeeding women
3. Medications: Beta blockers, corticosteroids, monoamine oxidase inhibitors, diabetes medications (including incretin mimetics and thiazolidinediones), and/or immunosuppressive therapy over the last 2 months.
4. Uncontrolled hypo- or hyperthyroidism
5. Current tobacco use
6. Active malignancy
7. History of clinically significant cardiac, hepatic, or renal disease.
8. History of any serious hypersensitivity reaction to study medications, any other incretin mimetic, any other formulation of supplemental vitamin B12, and/or cobalt
9. Personal or family history of Leber hereditary optic nerve atrophy
10. Prisoners or subjects who are involuntarily incarcerated
11. Compulsorily detention for treatment of either a psychiatric or physical (e.g., infectious disease) illness
12. Prior history of pancreatitis, medullary thyroid cancer, or multiple endocrine neoplasia type 2 (MEN 2)
13. Serum vitamin B12 level above the upper limit of assay detection

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2023-10-06 (Actual); Study Completion 2023-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Absalon D Gutierrez, MD, Principal Investigator — The University of Texas Health Science Center at Houston, Dept. of Medicine
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share all participant data (which will be deidentified) regarding our plasma samples, subcutaneous adipose tissue samples, and peripheral blood mononuclear cells. A study protocol and statistical analysis plan will be available as specified per policy of clinicaltrials.gov.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available one year after the primary completion date of the clinical trial, or 6 months post-publication, or 18 months after award end date - whichever comes first. Data will then be available indefinitely.
Access Criteria: Anyone can access the data via clinicaltrials.gov. If applicable, data will also be shared via the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) Information Network.

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (6 Weeks)
Arm/Group | Cyanocobalamin, Then Dulaglutide | Dulaglutide, Then Cyanocobalamin
Started | 17 | 6
Received Intervention | 16 | 6
Completed | 12 | 6
Not Completed | 5 | 0
Period: Washout (3 Weeks)
Arm/Group | Cyanocobalamin, Then Dulaglutide | Dulaglutide, Then Cyanocobalamin
Started | 12 | 6
Completed | 12 | 6
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Cyanocobalamin, Then Dulaglutide | Dulaglutide, Then Cyanocobalamin
Started | 12 | 6
Received Intervention | 12 | 6
Completed | 11 | 4
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyanocobalamin, Then Dulaglutide | Dulaglutide, Then Cyanocobalamin | Total
Number analyzed (Participants) | 17 | 6 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (7) | 39 (5) | 39 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 14
  Male | 8 | 1 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 1 | 2
  Black | 5 | 3 | 8
  Hispanic | 8 | 0 | 8
  Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 17 | 6 | 23
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 30.5 (3.4) | 31.4 (2.8) | 30.73 (3.26)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 126 (13) | 118 (11) | 123 (12)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters of mercury] | 79 (6) | 75 (8) | 77 (6)
Fasting Glucose Level [Mean (Standard Deviation); unit: milligrams per deciliter] | 94 (16) | 96 (14) | 94 (15)
percentage of glycosylated hemoglobin [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin"] | 5.5 (0.3) | 5.7 (0.1) | 5.5 (0.2)
Triglycerides Level [Mean (Standard Deviation); unit: milligrams per deciliter] | 135 (93) | 124 (86) | 132 (91)
Total Cholesterol Level [Mean (Standard Deviation); unit: milligrams per deciliter] | 193 (38) | 201 (31) | 195 (36)
high-density lipoprotein (HDL) Cholesterol Level [Mean (Standard Deviation); unit: milligrams per deciliter] | 56 (24) | 55 (8) | 55 (21)
low-density lipoprotein (LDL) Cholesterol Level [Mean (Standard Deviation); unit: milligrams per deciliter] | 111 (35) | 122 (28) | 113 (33)
aspartate aminotransferase (AST) Level [Mean (Standard Deviation); unit: units per liter] | 22 (8) | 19 (5) | 21 (7)
alanine aminotransferase (ALT) Level [Mean (Standard Deviation); unit: units per liter] | 24 (14) | 20 (10) | 22 (13)
Creatinine Level [Mean (Standard Deviation); unit: milligrams per deciliter] | 0.9 (0.3) | 0.9 (0.2) | 0.9 (0.2)
Hemoglobin Level [Mean (Standard Deviation); unit: grams per deciliter] | 14 (2) | 13 (2) | 13 (2)
Platelets Count [Mean (Standard Deviation); unit: billion cells per liter] | 296 (90) | 285 (51) | 293 (82)
thyroid-stimulating hormone (TSH) level [Mean (Standard Deviation); unit: milli-international units per liter] | 1.8 (1.4) | 1.8 (0.7) | 1.8 (1.2)
Vitamin B12 Level [Mean (Standard Deviation); unit: picograms per milliliter] | 497 (178) | 495 (255) | 496 (199)

OUTCOME MEASURES:

1. Primary Outcome: Cytokine Interleukin-6 (IL-6) Messenger Ribonucleic Acid (mRNA) Level (From Adipose Tissue)
Description: natural log transformed data is reported
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: natural log(arbitrary units)
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
natural log(arbitrary units) | 7.88 [7.16 to 8.60] | 7.67 [6.98 to 8.35]

2. Primary Outcome: Uncoupling Protein 1 (UCP1) Messenger Ribonucleic Acid (mRNA) Level (From Adipose Tissue)
Description: Uncoupling protein 1 (UCP1) is a marker of beige/brown fat. natural log transformed data is reported
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: natural log(arbitrary units)
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
natural log(arbitrary units) | 1.69 [-1.26 to 4.63] | 3.78 [1.68 to 5.87]

3. Primary Outcome: Signal Transducer and Activator of Transcription 3 (STAT3) Band Intensity/Western Blot (From Adipose Tissue)
Description: signaling intermediary with interleukin-6
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: PR Domain Containing 16 (PRDM16) Messenger Ribonucleic Acid (mRNA) Level ((From Adipose Tissue)
Description: PR domain containing 16 (PRDM16) is a marker of beige/brown fat. natural log transformed data is reported.
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: natural log(arbitrary units)
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
natural log(arbitrary units) | 2.58 [1.47 to 3.69] | 2.53 [1.48 to 3.58]

5. Secondary Outcome: Nicotinamide Adenine Dinucleotide Dehydrogenase (Ubiquinone) Iron-sulfur protein3 (NDUFS3) (From Adipose Tissue)
Description: marker of beige/brown fat
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Beta1-adrenoceptor (ADRB1) (From Adipose Tissue)
Description: marker of beige/brown fat
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Beta2-adrenoceptor (ADRB2) (From Adipose Tissue)
Description: marker of beige/brown fat
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Beta3-adrenoceptor (ADRB3) (From Adipose Tissue)
Description: marker of beige/brown fat
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Nuclear Factor Kappa B (NfKappaB) p65 Band Intensity/Western Blot (From Peripheral Blood Mononuclear Cells)
Description: signaling intermediary with interleukin-6
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Interleukin-6 (IL-6) mRNA (From Peripheral Blood Mononuclear Cells)
Description: cytokine
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: IL-6 (From Peripheral Blood Mononuclear Cells)
Description: cytokine
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Suppressor of Cytokine Signaling 3 (SOCS3) Band Intensity/Western Blot (From Peripheral Blood Mononuclear Cells)
Description: signaling intermediary with interleukin-6
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Cytokine IL-6 Level (From Plasma)
Description: natural log transformed data is reported.
  The "Measure Type" indicated as "Mean" actually refers to a "Adjusted Mean." Mean was adjusted for meteorological season. The meteorological season (i.e., spring, summer, fall, and winter) was adjusted for in the multivariable analysis as a potential confounding factor, since imbalances in ambient temperature between study arms could affect the findings.
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: natural log(picograms per milliliter)
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
natural log(picograms per milliliter) | -0.20 [-0.93 to 0.53] | -0.46 [-1.15 to 0.22]

14. Secondary Outcome: Free Fatty Acids Level (From Plasma)
Description: Free fatty acids level is a marker for insulin resistance. natural log transformed data is reported
  The "Measure Type" indicated as "Mean" actually refers to a "Adjusted Mean." Mean was adjusted for meteorological season. The meteorological season (i.e., spring, summer, fall, and winter) was adjusted for in the multivariable analysis as a potential confounding factor, since imbalances in ambient temperature between study arms could affect the findings.
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: natural log(nanomoles per liter)
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
natural log(nanomoles per liter) | -5.15 [-5.76 to -4.55] | -5.68 [-6.22 to -5.14]

15. Secondary Outcome: Insulin Level (From Plasma)
Description: Insulin Level is a marker of insulin resistance. natural log transformed data is reported.
  The "Measure Type" indicated as "Mean" actually refers to a "Adjusted Mean." Mean was adjusted for meteorological season. The meteorological season (i.e., spring, summer, fall, and winter) was adjusted for in the multivariable analysis as a potential confounding factor, since imbalances in ambient temperature between study arms could affect the findings.
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: natural log(picomoles per liter)
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
natural log(picomoles per liter) | 4.10 [3.77 to 4.43] | 3.86 [3.55 to 4.16]

16. Secondary Outcome: Glucose Level (From Plasma)
Description: Glucose Level is a marker of insulin resistance. The "Measure Type" indicated as "Mean" actually refers to a "Adjusted Mean." Mean was adjusted for meteorological season. The meteorological season (i.e., spring, summer, fall, and winter) was adjusted for in the multivariable analysis as a potential confounding factor, since imbalances in ambient temperature between study arms could affect the findings.
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: milligrams per deciliter
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
milligrams per deciliter | 80.61 [76.08 to 85.14] | 78.50 [74.22 to 82.78]

17. Secondary Outcome: Tumor Necrosis Factor - Alpha (From Plasma)
Description: as for outcome 13
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: natural log(picograms per milliliter)
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
natural log(picograms per milliliter) | .11 [-1.22 to 1.45] | 0.33 [-0.28 to 0.95]

18. Secondary Outcome: Interleukin-4 (From Plasma)
Description: cytokine
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Interleukin-10 (From Plasma)
Description: cytokine
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Interleukin-11 (From Plasma)
Description: cytokine
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Interleukin-13 (From Plasma)
Description: cytokine
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Glucagon-like Peptide-1 (From Plasma)
Description: The "Measure Type" indicated as "Mean" actually refers to a "Adjusted Mean." Mean was adjusted for meteorological season. The meteorological season (i.e., spring, summer, fall, and winter) was adjusted for in the multivariable analysis as a potential confounding factor, since imbalances in ambient temperature between study arms could affect the findings.
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: picomoles per milliliter
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
picomoles per milliliter | 40.66 [20.82 to 60.49] | 206.15 [187.42 to 224.88]

23. Secondary Outcome: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) is a marker of insulin resistance, calculated according to the formula: fasting insulin (mU/mL) x fasting glucose (mmol/L)/22.5 The "Measure Type" indicated as "Mean" actually refers to a "Adjusted Mean." Mean was adjusted for meteorological season. The meteorological season (i.e., spring, summer, fall, and winter) was adjusted for in the multivariable analysis as a potential confounding factor, since imbalances in ambient temperature between study arms could affect the findings.
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: HOMA-IR score
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
HOMA-IR score | 2.36 [1.77 to 2.95] | 1.63 [1.08 to 2.17]

24. Secondary Outcome: Fat Browning Measured as Standard Uptake Value (From Positron Emission Tomography - Computed Tomography (PET-CT) Reading)
Description: as for outcome 22
Time Frame: 6 weeks after start of each intervention
Measure: Mean (95% Confidence Interval); unit: standard uptake value
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 18 | 18
standard uptake value
  Right side PET- CT | 0.88 [0.23 to 1.52] | 1.37 [0.48 to 2.27]
  Left side PET-CT | 0.81 [0.23 to 1.39] | 1.26 [0.45 to 2.08]

25. Secondary Outcome: Oroboros Oxygen Consumption
Description: measure of oxygen consumption
Time Frame: 6 weeks after start of each intervention
Population: Data were not collected for this outcome measure.
Arm/Group | Cyanocobalamin | Dulaglutide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 17 weeks
Arm/Group | Cyanocobalamin | Dulaglutide
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1/23 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyanocobalamin (N=23) | Dulaglutide (N=23)
vasovagal response (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT04387201/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/01/NCT04387201/ICF_002.pdf